CLINICAL TRIAL: NCT02811601
Title: A Prospective Study of Port Site Pain Following Percutaneous Externally-Assembled Laparoscopic Urologic Surgery
Brief Title: Percutaneous Externally-Assembled Laparoscopic Urologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5160133
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Urologic Diseases
Keywords: Minimally Invasive Surgical Procedures
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEAL surgery (Experimental): Patients will undergo percutaneous externally-assembled laparoscopic surgery
  Interventions: Procedure: PEAL surgery

INTERVENTIONS:
Procedure: PEAL surgery — Patients will undergo percutaneous externally-assembled laparoscopic surgery where one or more 3 mm instruments are added or substituted for conventional 5 or 10 mm trocars.
  Other Names: PERCUTANEOUS EXTERNALLY-ASSEMBLED LAPAROSCOPIC (PEAL)

SUMMARY:
This will be a single-arm prospective internally-controlled study. Patients will undergo percutaneous externally-assembled laparoscopic surgery where one or more 3 mm instruments are added or substituted for conventional 5 or 10 mm trocars.

DETAILED DESCRIPTION:
The investigators have previously published a study regarding the use of a new surgical paradigm (percutaneous externally assembled laparoscopy, or PEAL) in porcine and cadaveric models in order to allow laparoscopic surgery to take place with improved cosmesis and decreased pain while still allowing the use of larger instruments and maintaining instrument triangulation. The investigators now seek to study the use of these instruments in the human patients undergoing laparoscopic urologic surgery.

This will be a single-arm prospective internally-controlled study. Patients will undergo percutaneous externally-assembled laparoscopic urologic surgery where one or more 3 mm instruments are added or substituted for conventional 5 or 10 mm trocars. Multiple outcome measures (endpoints) will be measured including time to first opioid use, total inpatient opioid dosage, patient ranking of painfulness of each port site, duration of ileus, time to ambulation, length of hospital stay, presence of any intraoperative or postoperative complications, operating time, estimated blood loss, and other routine parameters collected in a prospective surgical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic urologic surgery

Exclusion Criteria:

* Patients unwilling to participate in the study
* Patients unfit for laparoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06; Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Time to first opioid use | up to 30 days postoperatively
Total inpatient opioid dosage | up to 30 days postoperatively
Pain score of all surgical sites | up to 3 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Keheila, MD, Study Director — Loma Linda University Medical Center
Locations (1):
- Loma Linda Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arenas JL, Alsyouf M, Jang M, Myklak K, Faaborg D, Khater N, Baldwin DD. Percutaneous Externally Assembled Laparoscopic Instruments: Creation of a New Surgical Paradigm. J Endourol. 2016 Apr;30(4):433-40. doi: 10.1089/end.2015.0240. Epub 2016 Feb 9. PMID 26732739
- [Background] Rossitto C, Gueli Alletti S, Costantini B, Fanfani F, Scambia G. Total Laparoscopic Hysterectomy With Percutaneous (Percuvance) Instruments: New Frontier of Minimally Invasive Gynecological Surgery. J Minim Invasive Gynecol. 2016 Jan;23(1):14-5. doi: 10.1016/j.jmig.2015.09.004. Epub 2015 Sep 18. PMID 26386388
- [Background] Chang J, Boules M, Rodriguez J, Kroh M. Minilaparoscopy with Interchangeable, Full 5-mm End Effectors: First Human Use of a New Minimally Invasive Operating Platform. J Laparoendosc Adv Surg Tech A. 2016 Jan;26(1):1-5. doi: 10.1089/lap.2015.0418. Epub 2015 Nov 30. PMID 26618278